CLINICAL TRIAL: NCT00246870
Title: PET Imaging of GABA Receptors in Succinic Semialdehyde Dehydrogenase Deficiency
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060022; 06-N-0022
Record Dates: First submitted 2005-10-29; First posted 2005-10-31 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-10-19

CONDITIONS: Succinic Semialdehyde Dehydrogenase Deficiency; SSADH Deficiency
Keywords: Seizures; Development; Pediatric; Benzodiazepine Receptors; Neurotransmission; Succinic Semialdehyde Dehydrogenase; Deficiency; SSADH Deficiency; Healthy Volunteer; HV
MeSH Terms: conditions — succinic semialdehyde dehydrogenase deficiency; Seizures

SUMMARY:
This study will use brain imaging to map brain cell receptors for a chemical called GABA, a chemical that inhibits the activities of nerve cells. The study includes patients with succinic semialdehyde dehydrogenase deficiency, or SSADH (a disorder in which an enzyme deficiency disrupts GABA metabolism), their parents, and healthy volunteers. SSADH deficiency causes various neurological and neuromuscular problems, including mild to severe mental retardation, delays in the acquisition of skills requiring the coordination of mental and physical activities (psychomotor retardation), delays in language and speech development, and other symptoms.

Healthy volunteers 18-55 years of age, patients with SSADH between 5 and 24 years of age, and parents of patients 18-55 years of age may be eligible for this study.

Participants undergo magnetic resonance imaging (MRI) and positron emission tomography (PET) scanning as follows:

Magnetic resonance imaging

MRI uses a magnetic field and radio waves to produce images of body tissues and organs. For this procedure, the subject lies on a table that is moved into the scanner (a narrow metal cylinder surrounded by a magnetic field) wearing earplugs to muffle loud knocking and thumping sounds that occur during the scanning process. Scanning time varies from 20 minutes to 3 hours, with most scans lasting between 45 and 90 minutes. Participants may be asked to lie still for up to 90 minutes at a time. In addition to standard MRI, participants may also have new types of MRI that may detect brain abnormalities when regular MRI is normal, such as diffusion tensor MRI and magnetic resonance spectroscopy. There are no noticeable differences from ordinary MRI scans.

Positron Emission Tomography

A catheter (plastic tube) is placed in a vein in the subject's wrist. The subject lies on a table with his or her head placed in the scanner. A mask, used to help keep the head still in the scanner, is placed over the head. The mask is not uncomfortable and has holes for the subject to see through. A radioactive compound called flumazenil is injected into a vein. The scan takes about 90 minutes.

Some children need to be sedated for PET or MRI scans. In these cases, chloral hydrate, a standard drug for pediatric diagnostic procedures, is used.

...

DETAILED DESCRIPTION:
Objective: To measure CNS GABA receptors and GABA levels in patients with succinic semialdehyde dehydrogenase (SSADH) deficiency, a severe pediatric neurotransmitter disease.

Study Population: The study will include children and young adult patients with the disorder, as well as parents of patients (obligate heterozygotes), and adult normal volunteers.

Design: this is a natural history study using neuroimaging techniques. We will perform 11C-flumazenil PET scans, and magnetic resonance spectroscopy (MRS). We will perform neurological examinations to obtain data on clinical manifestations of the condition.

Outcome measures: The outcome measures will be the distribution of CNS binding of 11C-flumazenil, and brain GABA levels measured by MRS, and their relation to clinical manifestations such as motor, speech, and language impairment, hypotonia, hyporreflexia, and seizures. We expect to show that patients with SSADH deficiency will have multifocal reductions in FMZ binding and increased brain GABA levels in a similar pattern.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients

* Clinical characteristics consistent with SSADH deficiency.
* Persistent 4-hydroxybutyric aciduria (gamma-hydroxybutyric aciduria)
* Documented leucocyte extract succinic semialdehyde dehydrogenase enzyme deficiency
* English-speaking (or the ability to understand English as a second language)
* Patients may be male or female.
* Female patients of child bearing potential will have a pregnancy test within 24 hours of the study to ensure that pregnant patients will not participate.
* During the study, woman of child bearing potential must use a reliable method of birth control.

Parents

-Parents of affected patients are, by definition, heterozygous carriers of mutations in the succinic semialdehyde dehydrogenase gene.

EXCLUSION CRITERIA:

* Neither patients nor healthy volunteers may suffer from mental or physical illness that would interfere with participation.
* Neither patients nor healthy volunteers may be pregnant or nursing
* Neither patients nor healthy volunteers may use alcohol or recreational drugs during the study
* Patients requiring treatment of drugs known to affect the GABAergic system, including vigabatrin.
* Patients who had seizure activity 24 hours prior to the study.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10-24; Study Completion 2010-10-19

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - National Institute of Neurological Disorders and Stroke (NINDS), 9000 Rockville, Bethesda, Maryland

REFERENCES:
- [Background] Akaboshi S, Hogema BM, Novelletto A, Malaspina P, Salomons GS, Maropoulos GD, Jakobs C, Grompe M, Gibson KM. Mutational spectrum of the succinate semialdehyde dehydrogenase (ALDH5A1) gene and functional analysis of 27 novel disease-causing mutations in patients with SSADH deficiency. Hum Mutat. 2003 Dec;22(6):442-50. doi: 10.1002/humu.10288. PMID 14635103
- [Background] Al-Essa MA, Bakheet SM, Patay ZJ, Powe JE, Ozand PT. Clinical, fluorine-18 labeled 2-fluoro-2-deoxyglucose positron emission tomography (FDG PET), MRI of the brain and biochemical observations in a patient with 4-hydroxybutyric aciduria; a progressive neurometabolic disease. Brain Dev. 2000 Mar;22(2):127-31. doi: 10.1016/s0387-7604(99)00121-7. PMID 10722966
- [Background] Arnold S, Berthele A, Drzezga A, Tolle TR, Weis S, Werhahn KJ, Henkel A, Yousry TA, Winkler PA, Bartenstein P, Noachtar S. Reduction of benzodiazepine receptor binding is related to the seizure onset zone in extratemporal focal cortical dysplasia. Epilepsia. 2000 Jul;41(7):818-24. doi: 10.1111/j.1528-1157.2000.tb00248.x. PMID 10897152